CLINICAL TRIAL: NCT05062447
Title: Adaptive and Maladaptive Emotions in Patients With Cancer: Identification of Indicators
Acronym: EMOCA
Status: Terminated | Type: Observational
Why Stopped: No extention of the deadline was possible anymore.
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: Dutch Cancer Society (Other)
Responsible Party: Principal Investigator, Prof. dr. Joost Dekker, Principal Investigator, Amsterdam UMC, location VUmc
Other Study IDs: NL72824.029.20
Record Dates: First submitted 2021-08-25; First posted 2021-09-30 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Adaptation, Emotional
Keywords: cancer; patients; emotions; psychosocial; care
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Adaptive emotions, non-metastatic disease: Participants who are categorized as having 'adaptive emotions' and have a non-metastatic disease
- Adaptive emotions, metastatic disease: Participants who are categorized as having 'adaptive emotions' and have a metastatic disease
- maladaptive emotions, non-metastatic disease: Participants who are categorized as having 'maladaptive emotions' and have a non-metastatic disease
- maladaptive emotions, metastatic disease: Participants who are categorized as having 'maladaptive emotions' and have a metastatic disease

SUMMARY:
Primary Objective: To identify indicators distinguishing between adaptive and maladaptive emotions in patients with cancer.

DETAILED DESCRIPTION:
Background of the study:

The occurrence of cancer constitutes a major stressor, leading to a wide range of emotions. Patients need support from relatives, friends and caregivers to deal with these emotions. Some patients need professional mental health care, in addition to support. Unfortunately, an accurate instrument to identify patients in need of professional mental health care is not available. This leads to important mismatches in the provision of care.

In the field of oncology, the concept of 'distress' is used to refer to emotions associated with cancer. Measurement instruments (e.g. Distress Thermometer) are used to identify patients with clinically relevant distress. This approach results in major inconsistencies.While approximately one in three patients scores above the cut-off for distress, only about one in ten patients accepts mental healthcare, while it is unclear how many need mental health care.

In the field of mental health, it is generally acknowledged that a distinction needs to be made between normal and adaptive emotions versus maladaptive and psychopathological emotions in response to a potentially traumatic event such as cancer. The concept of distress fails to make this distinction. Some patients scoring above the cut-off for distress may indeed experience maladaptive emotions. Other patients scoring above the cut-off may actually experience adaptive emotions, which facilitate coping with cancer. Therefore, in order to provide appropriate care, identification of indicators distinguishing between adaptive and maladaptive emotions in patients with cancer is an urgent research priority.

Objective of the study:

To identify indicators that distinguish between adaptive and maladaptive emotions in patients with cancer, derived from recent innovative developments in the field of mental health.

Study design:

Patients are categorized as having 'adaptive emotions' or 'maladaptive emotions', using a reference standard: (a) a diagnostic mental health interview and questionnaires, or (b) patient's subjective need for professional mental health care. In all patients, emotional symptoms, cancer-treatment related symptoms and activities are assessed during a period of two weeks via mobile phone. Assessments of patients takes place twice; at 3 and 6 months after the start of chemo-or immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of a solid malignancy cancer, (i) non-metastatic disease or (ii) metastatic disease;
* between 3 and 7 months after start of treatment with (neo)adjuvant or 1st line chemotherapy or with (neo)adjuvant or 1st line immunotherapy;
* life expectancy of more than 3 months.

Exclusion Criteria:

* age < 18;
* insufficient command of the Dutch language;
* severe psychopathology, other than mood or anxiety disorder (e.g. lifetime history of bipolar disorder, schizophrenia, MDD (Major Depressive Disorder) with psychotic features, schizoaffective disorders);
* severe cognitive impairments (e.g. dementia);
* patients with a (indication of) brain tumor or -metastases;
* a history of severe drug or alcohol abuse within past 6 months;
* not competent in the use of a mobile phone
* no informed consent.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with solid malignancy, either (i) non-metastatic disease or (ii) metastatic disease, except for patients with a (indication of) brain tumor or -metastases. In each stratum (non-metastatic or metastatic disease), 40 patients with adaptive emotions and 40 patients with maladaptive emotions are recruited from the outpatient clinics at the Departments of Medical Oncology at seven major hospitals (160 patients in total). Patients are stratified by sex (female/male) and age (18-40; 40-70 and > 70 years old).
Sampling Method: Non-Probability Sample
Enrollment: 134 (Actual)
Dates: Start 2021-08-10 (Actual); Primary Completion 2024-05-06 (Actual); Study Completion 2024-05-06 (Actual)

PRIMARY OUTCOMES:
Emotional symptoms | During two weeks, once as soon as possible after inclusion and once three months later
  Prompted by Ecological Momentary Assessment (EMA), patients rate the following 15 mood states on a 7-point scale ranging from 1 'not at all' to 7 'very' (in the present study, we use 'emotional symptoms' to refer to these mood states). Emotional symptoms with a negative valence: feeling agitated, upset, irritated, listless/apathetic, down, nervous, bored, anxious, and worried. Emotional symptoms with a positive valence: satisfied, relaxed, cheerful, energetic, enthusiastic and calm. These items have been derived from the The Netherlands Study of Depression and Anxiety (NESDA) EMA diary-protocol, have sufficient with-in person variability and have been extensively used in previous studies.
Cancer-treatment-related symptoms | During two weeks, once as soon as possible after inclusion and once three months after first assessment
  Prompted by Ecological Momentary Assessment, patients rate the following six symptoms related to cancer-treatment on a 7-point scale ranging from 1 'not at all' to 7 'very': feeling tired, difficulty concentrating, nauseousness, loss of appetite, pain, and shortness of breath. These symptoms have been derived from the European Organisation For Research And Treatment Of Cancer (EORTC) item bank.
Activities related to the pursuit of life goals | During two weeks, once as soon as possible after inclusion and once three months after first assessment
  Prompted by Ecological Momentary Assessment, patients indicate whether they have been involved in the following five categories of activities: (a) work/study, (b) health-related activities (we will differentiate between activities focused on disease and treatment and activities focused on improving/maintaining physical fitness, and building or maintaining a healthy lifestyle), (c) social activities with relatives or friends, (d) intellectual and religious/spiritual activities, and (e) leisure/pleasure related activities.This question covers activities in the interval since the last assessment. The list of activities corresponds to the list of life goals (see below). Patients indicate in which activities they were involved. Combined with the patient's rating of the personal relevance of life goals (see below), this results in a rating of the involvement in specific activities related to the pursuit of personally relevant life goals.
Specific signs and symptoms as identified by oncologists and nurses | Once as soon as possible after inclusion in the study and once three months after first assessment
  In a qualitative study prior to this study, we have developed a checklist of potential signs and symptoms (e.g. a specific observation by an oncologist and nurse, such as crying or nervousness) which lead oncologists and nurses to suspect the need for professional mental health care among their patients. This checklist will be filled in by an oncologist and a nurse.
Life goals | Once as soon as possible after inclusion in the study and once three months after first assessment
  Patients are interviewed about their life goals. In the interview, they are presented with an empirically-derived list of potential life goals, in five categories: (a) achievement or work/study related goals, (b) health-related goals (we will differentiate between goals focused on disease and treatment and goals focused on improving/maintaining physical fitness, and building or maintaining a healthy lifestyle), (c) social goals, (d) psychological goals that focus on inner psychological states, and (e) leisure/pleasure related goals (cheerfulness/fun). Subsequently, patients assess to what extent they are striving to attain these goals, on a 5-point Likert scale raging from 1 'not at all' to 5 'very' (i.e. they rate the personal relevance of these life goals). The scores are used to weigh the five categories of activities (see above).
Diagnostic mental health interview | Once as soon as possible after inclusion in the study and once three months after first assessment
  The Composite International Diagnostic Interview (CIDI) (version 2.1) is a comprehensive, fully-structured interview for the assessment of lifetime and current (1 month recency) mental disorders, used to assess the presence of depression and anxiety disorder. In addition, we use the Four-dimensional symptom questionnaire (4DSQ) (Vier Dimensionele Klachten Lijst (4DKL) to assess adjustment disorder, with patients scoring > 20 on Distress and without a depressive or anxiety disorder on the CIDI categorized as having an adjustment disorder. The interview is conducted in person by a well-trained researcher. Maladaptive emotions are rated as present if the patient scores positive on major depressive disorder, an anxiety disorder (panic disorder, agoraphobia without panic, specific phobia, social phobia, generalized anxiety disorder, and posttraumatic stress disorder) or adjustment disorder.
The need for professional mental health care | Once as soon as possible after inclusion in the study and once three months after first assessment
  The Distress Thermometer is a single item self-report measure of distress. Patients are asked to rate their overall distress on a visual scale from 0 (no distress) to 10 (extreme distress). The Problem List identifies problems in five domains: the practical, social, cognitive-emotional, spiritual/religious and physical domain. Patients indicate whether in the last three months they experienced a problem in these domains, using a five-point scale (ranging from 1 'no problem at all' to 5 'very much a problem'). For every domain in which patients report at least one problem, we ask whether they (a) received a referral for the problem, (b) did not receive a referral, but would have preferred a referral for the problem, (c) did not want or receive a referral for the problem, but would be willing to consider a referral in the future, or (d) did not want or receive a referral, neither in the present nor the future.
Threatening experiences | Once as soon as possible after inclusion in the study and once three months after first assessment
  The List of Threatening Experiences is a brief life events questionnaire, assessing the occurrence of 12 events (never, past year, life time)

SECONDARY OUTCOMES:
Pittsburgh Sleep Quality Index | Once as soon as possible after inclusion in the study and once three months after first assessment
  Pittsburgh Sleep Quality Index is a 19 item self-report questionnaire assessing sleep quality and quantity. There are 7 component scores: subjective sleep quality, sleep latency, duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction
Mastery | Once as soon as possible after inclusion in the study and once three months after first assessment
  Mastery is the feeling to which a person perceives himself or herself to be in control of events and ongoing situations. The 5-item abbreviated mastery scale will be used. A 5-point Likert scale is used to rate each item (e.g. 0 = strongly disagree, 4 = strongly agree).
Emotional reactivity in daily life | Once as soon as possible after inclusion in the study and once three months after first assessment
  Participants are asked whether they agree, disagree or are unsure about 3 statements concerning emotional reactivity in daily life (e.g. "Sometimes my feelings are strong, but they don't get in the way of day to day life), and how often (always, often, sometimes, rarely, never) 2 situations concerning emotional reactivity in daily life occur (e.g. How often do you find that your emotions are very unstable, or swing from one extreme to another in a way you sometimes find hard to control?).
Social and instrumental support | Once as soon as possible after inclusion in the study and once three months after first assessment
  The Close Person Inventory is a 14 item self-report questionnaire that will be used to measure social support received from the individual reported as being closest to the participant during the previous 12-month period. A 5-point Likert scale is used to measure how often they experience 3 components of social support: confiding/emotional, practical and negative social support (0 = never, 4 = very often).

CONTACTS AND LOCATIONS:
Overall Officials: Prof. dr. J. Dekker, Principal Investigator — VUmc
Locations (6):
- Netherlands (6):
  - VU University Medical Center, Amsterdam, North Holland
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch
  - Rijnstate, Arnhem
  - Slingeland Ziekenhuis, Doetinchem
  - Radboud UMC, Nijmegen
  - Isala Klinieken Zwolle, Zwolle

IPD SHARING:
Plan to Share IPD: No